CLINICAL TRIAL: NCT03608345
Title: Effects of Space Maintainers on Oral Health
Brief Title: Effects of Fixed and Removable Space Maintainers on Periodontal Health and DMFT/Dft Values
Status: Completed | Type: Observational
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Aliye Tugce Gurcan, Assist. Prof., Altinbas University
Other Study IDs: Altinbas University
Record Dates: First submitted 2018-07-02; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Dental Plaque
Keywords: oral health; dental plaque; space maintenance
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: space maintainer — Space maintainers are applied after the missing teeth in pediatric dentistry for protection of size of extracted area.

SUMMARY:
Space maintainers are appliances that applied when primary teeth were lost prematurely because of many reasons such as tooth decay, trauma, lack of germ of permanent tooth.4 Space problems play an important role in practice of dentistry and also understanding of the dental development in the primary and mixed dentitions could help to intercept the malocclusion.The aim of this study is to evaluate the effects of applied space maintainers on periodontal health and dental status after teeth missing in pediatric dentistry clinic.

DETAILED DESCRIPTION:
The study was approved by the Ethics Committee of the Istanbul University Faculty of Dentistry (No:2014/8) and was carried out in agreement with the Declaration of Helsinki principles. This study conducted 104 patient whose age between the range of 4-15 years were chosen to applied fixed (band and loop, palatal arch, lingual arch) or removable space maintainers in Istanbul University Faculty of Dentistry Department of Pediatric Dentistry were followed between years of 2013-2014. Totally, four of the patients excluded due to systemically and genetically disorder.

In primary and mixed dentition, dft index was used and in permanent dentition DMFT index was used. Longevity time in the mouth, the number of developing new caries were evaluated and DMFT/dft and plaque index were compared.

ELIGIBILITY:
Inclusion Criteria:

* healthy and applied space maintainer patients

Exclusion Criteria:

* unhealthy and non-applied space maintainer patients

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 100 patient whose age between a range of 4-15 years due to having early loss of teeth and were treated with fixed and removable space maintainers in Istanbul University Faculty of Dentistry Department of Pediatric Dentistry were included to this study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
DMFT/dft index value changes after applying space maintainers | 12 months
  With visual examination DMFT/dft index value changes were recorded to patient files

SECONDARY OUTCOMES:
Plaque index value changes after applying space maintainers | 12 months
  With visual examination and rounded explorer, plaque index value changes were recorded to patient files according to Sillness and Loe.

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Tuğçe Gürcan, Assist.Prof., Principal Investigator — Altinbas University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arikan V, Kizilci E, Ozalp N, Ozcelik B. Effects of Fixed and Removable Space Maintainers on Plaque Accumulation, Periodontal Health, Candidal and Enterococcus Faecalis Carriage. Med Princ Pract. 2015;24(4):311-7. doi: 10.1159/000430787. Epub 2015 Jun 4. PMID 26044443
- [Background] American Academy on Pediatric Dentistry Clinical Affairs Committee-Developing Dentition Subcommittee; American Academy on Pediatric Dentistry Council on Clinical Affairs. Guideline on management of the developing dentition and occlusion in pediatric dentistry. Pediatr Dent. 2008-2009;30(7 Suppl):184-95. No abstract available. PMID 19216419
- [Background] Arikan F, Eronat N, Candan U, Boyacioglu H. Periodontal conditions associated with space maintainers following two different dental health education techniques. J Clin Pediatr Dent. 2007 Summer;31(4):229-34. doi: 10.17796/jcpd.31.4.9588m43n027t560n. PMID 19161056